CLINICAL TRIAL: NCT01644370
Title: Allergen Specific T Effector and T Regulatory Cell Response to Common Aeroallergens Following Immune Restoration in HIV-infected Children
Brief Title: Children With HIV and Asthma (CHIVAS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The HIV Netherlands Australia Thailand Research Collaboration (Other)
Collaborators: Chulalongkorn University (Other); National Health Security Office, Thailand (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: HIV-NAT 102
Record Dates: First submitted 2012-07-17; First posted 2012-07-19 (Estimated); Last update posted 2016-02-22 (Estimated); Status verified 2016-02

CONDITIONS: T Cell Response to Asthma in HIV-infected Patients Before and After Starting Treatment
Keywords: HIV-infected children; T cell response; asthma
MeSH Terms: conditions — Asthma | interventions — Antiretroviral Therapy, Highly Active

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- HIV positive with aeroallergen (Other): positive for aeroallergen at baseline
  Interventions: Drug: HAART
- HIV positive without aeroallergen (Other): negative for aeroallergen at baseline
  Interventions: Drug: HAART
- control (No Intervention): HIV negative children (n=10)

INTERVENTIONS:
Drug: HAART — as per Thai HIV Treatment guidelines
  Arms: HIV positive with aeroallergen; HIV positive without aeroallergen

SUMMARY:
To explore allergen-specific effector and regulatory T cell response in HIV-infected children before and after HAART initiation

DETAILED DESCRIPTION:
Recently, US investigators have observed that HIV-infected (HIV+) children on highly active antiretroviral therapy (HAART) have a much greater cumulative incidence of asthma.Regulatory T cells may mitigate the pathogenicity of asthma through the suppression of Th2 responses. Since asthma is predominantly a TH2 mediated condition, we propose that new onset of asthma after HAART in HIV- infected children may be secondary to dysregulated immune reconstitution. The restoration of CD4+ T cell-mediated immunity in HIV+ patients treated with HAART may lead to airway inflammation, narrowing, hyperresponsiveness, and possibly remodeling.

The increased incidence of asthma in HIV-infected children treated with HAART is likely secondary to multiple factors that may include hypersensitivity to certain aeroallergens, dysregulation of effector and regulatory T cell response, as well as the imbalance of TH1 vs. TH2 cytokines. Therefore this study will identify the immunopathogenesis of increased airway hyperresponsiveness in HIV-positive patients.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 2-18 years
2. Parent signed inform consent and children signed assent form
3. Children who are starting highly active antiretroviral therapy (HAART) due to clinical indication or switching HAART due to treatment failure within 45 days after screening visit

Exclusion Criteria:

1. Pregnancy
2. History of chronic lung disease including lymphoid interstitial pneumonitis (LIP), and bronchopulmonary dysplasia (BPD).
3. Active opportunistic infections i.e. pulmonary tuberculosis, PCP, pneumonia
4. Conditions limiting ability of subject to comprehend questionnaires (i.e. mental retardation).

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2011-09; Primary Completion 2014-07 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
T cell response | 24 weeks
  exploring T cell response by immunophenotyping and cytokine detection in HIV-infected children before and after HAART initiation

CONTACTS AND LOCATIONS:
Overall Officials: Praphan Phanuphak, MD, PhD, Principal Investigator — The HIV Netherlands Australia Thailand Research Collaboration
Locations (2):
- Thailand (2):
  - The HIV Netherlands Australia Thailand Research Collaboration (HIV-NAT), Bangkok
  - The King Chulalongkorn Memorial Hospital, Chulalongkorn University, Division of Allergy & Immunology, Department of Pediatrics, Bangkok

REFERENCES:
- See also: HIV Netherlands Australia Thailand Research Collaboration (HIV-NAT) — http://www.hivnat.org